CLINICAL TRIAL: NCT01385527
Title: Using an Internet Survey to Improve Adherence in Pediatric Atopic Dermatitis
Brief Title: Pediatric Atopic Dermatitis (AD) Internet Survey
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study was never initiated, No participants enrolled
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IRB00016545
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weekly Internet survey w medication (Experimental): Weekly survey via email plus topical triamcinolone
  Interventions: Behavioral: Weekly Internet survey; Drug: Topical Triamcinolone
- Topical triamcinolone only (Active Comparator): Standard of care
  Interventions: Drug: Topical Triamcinolone

INTERVENTIONS:
Behavioral: Weekly Internet survey — Parents will complete a weekly online survey about medication use.
  Arms: Weekly Internet survey w medication
Drug: Topical Triamcinolone — Topical triamcinolone to all affected areas once daily

SUMMARY:
The purpose of this study is to evaluate whether participation in an Internet-based intervention helps improve atopic dermatitis treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any child age 2 to 8 with a diagnosis of atopic dermatitis confirmed by a dermatologist, together with the child's parent/guardian. Written consent must be given by parent/guardian.

Exclusion Criteria:

* Child is less than 2 or greater than 8 years of age.
* Known allergy or sensitivity to topical triamcinolone in the child.
* Inability to complete all study-related visits, or inability to complete the Internet survey due to inadequate Internet access.
* Introduction of any other prescription medication, topical or systemic, for atopic dermatitis while participating in the study. Subjects who are on systemic anti-inflammatory treatments for atopic dermatitis must be on a stable dose for at least 3 months prior to enrollment.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2014-10-27 (Actual); Study Completion 2014-10-27 (Actual)

PRIMARY OUTCOMES:
Adherence to topical triamcinolone | 12 weeks

SECONDARY OUTCOMES:
Eczema Area Severity Index | 12 weeks
Investigator's Global Assessment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No